CLINICAL TRIAL: NCT00536835
Title: A Phase I Study to Determine the Safety, Pharmacokinetics, and Pharmacodynamics of [GSK461364], a Polo-like Kinase 1 (PLK1) Inhibitor, in Adult Subjects With Advanced Solid Tumor or Non-Hodgkins Lymphoma
Brief Title: Study to Assess the Pharmacokinetics and Pharmacodynamics of GSK461364 in Subjects With Non-Hodgkins Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLK107427
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2017-06-26 (Actual); Status verified 2017-06

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkins Lymphoma; Cancer; First time in human; PLK1 inhibitor; Advanced Solid Tumor; GSK461364
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — GSK 461364

ARMS (2):
- Stage A (Experimental): Stage A will identify maximum tolerated doses for either Schedule 1 - GSK461364 given once weekly on Day 1, 8 and 15 every 28 days; Schedule 2 - GSK 461364 given twice weekly Days 1, 2, 8, 9, 15 and 16; Schedule 3 Daily on Day 1 to Day 15 every 21 days.
  Interventions: Drug: GSK461364
- Stage B (Experimental): Evaluate safety, PK, pharmacodynamic (PD) & tumor response in expanded cohorts at the MTD for at least one schedule from Stage A.
  Interventions: Drug: GSK461364

INTERVENTIONS:
Drug: GSK461364 — GSK461364 will be given intravenously as a 4 hour infusion in either a final volume of 500 or 1000 mLs. The starting dose for Stage A - Schedule 1 was 50 mg and doses were to be escalated as described in protocol until maximum tolerated dose established.

SUMMARY:
This is a first time in human study that is being done to determine the maximum tolerated dose and initial pharmacokinetic parameters of GSK461364, given by IV, in adult subjects with solid tumors and Non-Hodgkins lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of advanced solid tumor or Non-Hodgkins Lymphoma (excluding HIV-associated lymphoma) that has relapsed or is refractory to standard therapies
* At least 18 years of age
* Female who are of non-childbearing potential or who have a negative pregnancy test who uses approved contraception
* Male with a female partner of childbearing potential must have had a vasectomy or both are using approved contraception
* Lab values that are within range as described in the protocol
* Paraffin-embedded archival tumor tissue available for testing
* Signed written informed consent

Exclusion Criteria:

* Undergone major surgery or received anti-cancer therapy
* History of hemolytic anemia
* Clinical lab tests that are out of range as described in the protocol
* Females who are pregnant or lactating
* Significant heart problems
* Serious or unstable pre-existing medical or psychiatric condition
* Are not able to comply with the study protocol
* Use of prohibited medications
* Have low blood pressure
* Evidence of symptomatic or untreated central nervous system involvement and require corticosteroids or anti-epileptic meds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08-16 (Actual); Primary Completion 2009-09-29 (Actual); Study Completion 2009-09-29 (Actual)

PRIMARY OUTCOMES:
Plasma levels for GSK461364 will be taken at:Schedule 1:Day 1, 8, 15, & 22 for Cycle 1 and Day 1, 8 & 15 for subsequent cycles.Schedule 2:Day 1, 2, 8, 9, 15, & 16 for all cycles.Schedule 3:Day 1 to 5 for all cycles. | 16 Days

SECONDARY OUTCOMES:
Safety will be evaluated by: - Physical exam at screen & then D1 for each cycle - 12 lead ECG & telemetry at screen & Wk 1 to 3 for Schedule 1 & 2, & Wk 1 & 2 (ECG only) for Schedule 3. - Lab tests & AE monitoring throughout the study. | 16 Days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United Kingdom (3):
  - GSK Investigational Site, Sutton, Surrey
  - GSK Investigational Site, Belfast, Northern Ireland
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Olmos D, Barker D, Sharma R, Brunetto AT, Yap TA, Taegtmeyer AB, Barriuso J, Medani H, Degenhardt YY, Allred AJ, Smith DA, Murray SC, Lampkin TA, Dar MM, Wilson R, de Bono JS, Blagden SP. Phase I study of GSK461364, a specific and competitive Polo-like kinase 1 inhibitor, in patients with advanced solid malignancies. Clin Cancer Res. 2011 May 15;17(10):3420-30. doi: 10.1158/1078-0432.CCR-10-2946. Epub 2011 Apr 1. PMID 21459796
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study 107427 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/PLK107427?search=study&study_ids=107427#rs
- Available data/document: Clinical Study Report: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: PLK107427 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register